CLINICAL TRIAL: NCT01838044
Title: A Randomized Double Blind Placebo Controlled Parallel Group Study Of The Efficacy And Safety Of Concomitant Administration Of Celecoxib And Pregabalin Compared With Celecoxib Monotherapy, In Patients With Chronic Low Back Pain Having A Neuropathic Component
Brief Title: Efficacy and Safety Study of Celecoxib and Pregabalin Compared With Celecoxib Monotherapy, in Patients With Chronic Low Back Pain Having a Neuropathic Component
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment terminated on 3Apr2015 due to slow recruitment rate and lack of operational feasibility. Study was not terminated for reasons of safety/efficacy.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081296
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2016-07

CONDITIONS: Chronic Low Back Pain With a Neuropathic Component
MeSH Terms: interventions — Pregabalin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): The group of patients who are randomized to receive concomitant treatment of pregabalin and celecoxib during the first study period.
  Interventions: Drug: pregabalin and celecoxib
- Arm B (Other): The group of patients who are randomized to receive celecoxib monotherapy during the first study period.
  Interventions: Drug: Placebo and celecoxib

INTERVENTIONS:
Drug: pregabalin and celecoxib — During the first study period subjects in Arm A will be administered a daily fixed dose of celecoxib 200 mg once daily and pregabalin 150 mg (75 mg BID) for one week (during Week 0) followed by pregabalin 300 mg (150 mg BID) daily for the remaining 4 weeks. During the second study period all subjects will be administered concomitant treatment of a daily fixed dose of celecoxib 200 mg once daily and pregabalin 300 mg (150 mg BID). Subjects in Arm B will be initiated on pregabalin 150 mg (75 mg BID) daily for one week, before pregabalin will up titrated to 300 mg (150 mg BID) daily.
  All subjects will complete a treatment taper (a) after completing the second study period or (b) after premature study discontinuation. During treatment taper, the pregabalin dose will be decreased to 150 mg (75 mg BID) daily and subjects will participate in a follow up visit for a final safety assessment.
  Arms: Arm A
Drug: Placebo and celecoxib — Subjects in Arm B will be administered a daily fixed dose celecoxib 200 mg and placebo of pregabalin for 5 weeks. During the second study period all subjects will be administered concomitant treatment of a daily fixed dose of celecoxib 200 mg once daily and pregabalin 300 mg (150 mg BID). Subjects in Arm B will be initiated on pregabalin 150 mg (75 mg BID) daily for one week, before pregabalin will up titrated to 300 mg (150 mg BID) daily.
  All subjects will complete a treatment taper (a) after completing the second study period or (b) after premature study discontinuation. During treatment taper, the pregabalin dose will be decreased to 150 mg (75 mg BID) daily and subjects will participate in a follow up visit for a final safety assessment.
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine if treatment with celecoxib and pregabalin together would prove to be more effective in relief of pain than treatment with celecoxib alone in people who have chronic low back pain with a probable neuropathic component.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of the concomitant use of pregabalin and celecoxib compared with celecoxib monotherapy for the symptomatic relief of pain in patients with chronic low back pain with a probable neuropathic component.

The secondary objectives are:

* Demonstrate the additional benefit of adding pregabalin to celecoxib monotherapy.
* To evaluate the concomitant use of pregabalin and celecoxib compared to celecoxib monotherapy in a set of patient reported measures (sleep, depression, anxiety, impact of pain in daily functions, patient's global impression of change and patient's perception of the treatment).
* To evaluate the safety and tolerability of celecoxib and of the concomitant administration of pregabalin and celecoxib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have Chronic low back pain with high probability of a significant neuropathic component for 4 years or less (but no less than 3 months)
* Subjects must be in generally good health, except for the presence of chronic low back pain with a neuropathic component.
* Subjects must be literate and have the ability (unaided) to understand and use the interactive voice response system (IVRS), have daily access to a telephone or the internet in order to complete the IVRS assessments each day, perform telephone or web visits and complete all required assessments/forms

Exclusion Criteria:

* Subjects with past history of surgery for chronic low back pain.
* Subjects with past history of failure on pregabalin treatment and/or intolerance associated with pregabalin or gabapentin.
* Subjects with past history of intolerance associated with celecoxib or known hypersensitivity to celecoxib.
* Patients with anticipated need for treatment with opioid analgesics, anti-epileptic medications, SNRI antidepressants or tricyclic antidepressants to alleviate pain during the course of the study.
* Patients with chronic low back pain with a neuropathic component for more than 4 years.
* Patients with neurologic disorders unrelated to low back pain that may confuse or confound the assessment of neuropathic pain (eg, primary or secondary nerve diseases).
* Subjects considered at risk of suicide or self-harm based on investigator judgment and/or details of a risk assessment.
* Use of prohibited medications in the absence of appropriate washout periods.
* Patients with any severe pain associated with conditions other than chronic low back pain with a neuropathic component that may confound the assessment or self-evaluation of the pain due to chronic low back pain.
* Patients with diabetes with poor glycemic control (HbA1c >8%).
* Patients with any clinically significant or unstable medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, would compromise participation in the study
* Patients who have participated in any previous clinical trial for pregabalin or have participated in 2 or more previous clinical trials for pain related to chronic low back pain.
* Patients who are likely to require surgery during the course of the study (except minor surgery, eg, for skin conditions)
* Patients with a history of Substance Abuse as defined by DSM-IV-TR diagnostic criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Brazil (7):
  - Centro de Pesquisa Clínica do Hospital Universitário da Universidade Federal do Maranhão - CEPEC, São Luís, Maranhão
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - CMIP-Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - EDUMED Educação em Saúde - Centro de Pesquisas Clínicas, Curitiba, Paraná
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto Paulista de Reumatologia da UNIFESP, São Paulo, São Paulo
  - Instituto de Pesquisa Clinica e Medicina Avancada - IMA Brasil, São Paulo
- Chile (2):
  - Centro de Diagnostico y Tratamiento Ltd. Clinica Siresa, Temuco, Región de la Araucanía
  - Centro de Investigación Clínica Neuropsicología Ltda, La Florida, Santiago Metropolitan
- Colombia (2):
  - Fundacion Cardiovascular de Colombia - Instituto del Corazon Floridablanca, Floridablanca, Santander Department
  - Centro Medico Imbanaco C.M.I (Sede 01 and Sede 02) / Sede 12 Centro Medico Imbanaco de Cali S.A., Santiago de Cali
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Umum Sarawak (Sarawak General Hospital), Kuching, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
- Mexico (10):
  - Centro Integral en Reumatología SA de CV, Guadalajara, Jalisco
  - Clinica De Investigacion En Reumatologia Y Obesidad S.C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica SC., Guadalajara, Jalisco
  - Hospital Angeles Chapalita, Guadalajara, Jalisco
  - Unidad de Cancerología, Zapopan, Jalisco
  - MENTRIALS S. A. de C. V., Mexico City, Mexico City
  - Accelerium S. de R.L de C.V., Monterrey, Nuevo León
  - Unidad de Atención Médica e Investigacion en salud, Mérida, Yucatán
  - Unidad de Atencion Medica e Investigación en salud SC, Mérida, Yucatán
  - Centro de Investigacion y Atencion Integral de Durango SC, Durango
- Raffles Hospital, Singapore, Singapore
- Thailand (3):
  - Maharaj Nakorn ChiangMai Hospital, Muang, Chiang Mai
  - Sappasithiprasong Hospital, Muang, Ubonratchathani Thailand
  - Division of Neurology ,, Bangkok

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081296&StudyName=Efficacy%20and%20Safety%20Study%20of%20Celecoxib%20and%20Pregabalin%20Compared%20with%20Celecoxib%20Monotherapy%2C%20in%20Patients%20with%20Chronic%20Low%20Back%20Pain%20Havi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 28 sites across 7 countries. From a total of 232 participants screened, 180 were randomized into Period 1 and 166 entered into Period 2.
Pre-assignment Details: Participants who completed a minimum of 4 days per week of daily diaries during the 7 days preceding the baseline visit and had a mean weekly pain score >= 4 at the end of screening were randomized to either Arm A or Arm B.
Groups:
- Arm A: During Period 1, participants in Arm A were administered a daily fixed dose of celecoxib 200 mg once daily and pregabalin 150 mg (75 mg twice-daily [BID]) for 1 week followed by pregabalin 300 mg (150 mg BID) daily for the remaining 4 weeks (during Weeks 2, 3, 4 and 5). During Period 2, all participants were administered concomitant treatment of a daily fixed dose of celecoxib 200 mg once daily and pregabalin 300 mg (150 mg BID). All participants completed a treatment taper (a) after completing the second study period or (b) after premature study discontinuation. During treatment taper, the pregabalin dose was decreased to 150 mg (75 mg BID) daily and participants had participated in a follow up visit for a final safety assessment.
- Arm B: During Period 1, participants in Arm B were administered a daily fixed dose of celecoxib 200 mg and placebo of pregabalin for 5 weeks (during Weeks 1, 2, 3, 4 and 5). During Period 2, all participants were administered concomitant treatment of a daily fixed dose of celecoxib 200 mg once daily and pregabalin 300 mg (150 mg BID). Participants in Arm B were initiated on pregabalin 150 mg (75 mg BID) daily for 1 week, before pregabalin was up-titrated to 300 mg (150 mg BID) daily. All participants completed a treatment taper (a) after completing the second study period or (b) after premature study discontinuation. During treatment taper, the pregabalin dose was decreased to 150 mg (75 mg BID) daily and participants had participated in a follow up visit for a final safety assessment.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 89 | 91
Completed | 81 | 75
Not Completed | 8 | 16
Not completed — Adverse Event | 4 | 6
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Insufficient clinical response | 1 | 2
Not completed — Medication error without associated AE | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population was composed of all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (11.7) | 49.2 (12.2) | 49.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Mean Pain Numeric Rating Scale (NRS) Score at Week 5 (ie, Visit 4) Compared Between the Two Study Arms
Description: The Daily Pain diary consists of an 11-point NRS ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10: Select the number that best describes your pain during the past 24 hours from 0 to10 where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: Baseline and Week 5
Population: The Full Analysis Set (FAS) that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale | -2.18 (0.212) | -2.03 (0.212)
Statistical Analysis 1: Comparison: Arm A vs Arm B; Statistical analysis at Week 5 compared between two study arms; Test type: Superiority or Other; p = 0.6012, Mixed Models Analysis; LS Mean Difference = -0.15, 95% CI 2-sided [-0.72 to 0.42], Standard Error of Mean 0.287

2. Secondary Outcome: Change in the Weekly Mean Pain NRS Score in Arm B, Compared Between Week 5 (Visit 4) and Week 10 (Visit 6).
Description: as for outcome 1
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm B
Number analyzed (Participants) | 91
Units on a scale | 1.42 (0.204)
Statistical Analysis 1: Comparison: Arm B; Statistical analysis of weekly mean pain NRS score in Arm B at Week 10; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [1.02 to 1.83]

3. Secondary Outcome: Change From Baseline in the Weekly Mean Pain NRS Score at Week 10 (Visit 6) Compared Between the Two Study Arms
Description: as for outcome 1
Time Frame: Baseline and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale | -3.21 (0.262) | -3.45 (0.265)
Statistical Analysis 1: Comparison: Arm A vs Arm B; Statistical analysis of weekly mean pain NRS score in Arm B compared between two study arms at Week 10; Test type: Superiority or Other; p = 0.5128, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.48 to 0.95], Standard Error of Mean 0.361

4. Secondary Outcome: Change From Baseline in Benefit, Satisfaction, and Willingness to Continue Measure Scores Compared Between Arms at Week 5 (Visit 4) and at Week 10 (Visit 6)
Description: The BSW consists of 3, single-item measures designed to capture the participant's perception of the effect of treatment in terms of the relative benefit, their satisfaction, and their intention or willingness to continue on therapy. The BSW was administered by the investigator or designated site personnel in the local language as a standardized interview during the follow-up visits. The BSW can potentially be self-administered; however, this method of administration has not been tested. Participants completed this questionnaire at Visit 4 and Visit 6.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Percentage of participants
  Benefit from Treatment - No benefit (Week 5) | 10.1 | 6.6
  Benefit from Treatment - Little benefit (Week 5) | 22.5 | 29.7
  Benefit from Treatment - Much benefit (Week 5) | 61.8 | 53.8
  Satisfaction from Treatment - DVN (Week 5) - Yes | 78.7 | 84.6
  Satisfaction from Treatment - DVN (Week 5) - No | 15.7 | 5.5
  A Little Satisfied (Week 5) | 20.2 | 26.4
  Very Satisfied (Week 5) | 58.4 | 58.2
  A Little Dissatisfied (Week 5) | 12.4 | 4.4
  Very Dissatisfied (Week 5) | 3.4 | 1.1
  Willingness to Continue - DVN (Week 5) - Yes | 94.4 | 89.0
  Willingness to Continue - DVN (Week 5) - No | 0 | 1.1
  A Little Bit Willing (Week 5) | 5.6 | 4.4
  Very Willing (Week 5) | 88.8 | 84.6
  A Little Unwilling (Week 5) | 0 | 0
  Very Unwilling (Week 5) | 0 | 1.1
  Benefit from Treatment - No benefit (Week 10) | 4.5 | 3.3
  Benefit from Treatment - Little benefit (Week 10) | 14.6 | 9.9
  Benefit from Treatment - Much benefit (Week 10) | 71.9 | 70.3
  Satisfaction from Treatment - DVN (Week 10) - Yes | 83.1 | 80.2
  Satisfaction from Treatment - DVN (Week 10) - No | 7.9 | 3.3
  A Little Satisfied (Week 10) | 9.0 | 11.0
  Very Satisfied (Week 10) | 74.2 | 69.2
  A Little Dissatisfied (Week 10) | 5.6 | 2.2
  Very Dissatisfied (Week 10) | 2.2 | 1.1
  Willingness to Continue - DVN (Week 10) - Yes | 88.8 | 81.3
  Willingness to Continue - DVN (Week 10) - No | 2.2 | 2.2
  A Little Bit Willing (Week 10) | 4.5 | 4.4
  Very Willing (Week 10) | 84.3 | 76.9
  A Little Unwilling (Week 10) | 0 | 0
  Very Unwilling (Week 10) | 2.2 | 2.2

5. Secondary Outcome: Patient Global Impression of Change (PGIC) Compared Between Arms at Week 5 (Visit 4) and at Week 10 (Visit 6)
Description: The PGIC is a single-item, self-rated instrument that measures change in the patient's overall status since starting study medication on a scale from 1 (very much improved) to 7 (very much worse), where lower scores indicate greater improvement. This scale was administered at Visit 4 and Visit 6.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5 (n=84, 82) | 2.69 (0.11) | 2.64 (0.11)
  Week 10 (n=81, 76) | 2.31 (0.10) | 2.11 (0.11)
Statistical Analysis 1: Comparison: Arm A vs Arm B; Statistical analysis at Week 5 based on comparison between treatment groups; Test type: Superiority or Other; p = 0.7251, Mixed Models Analysis; LS Mean Difference = 0.05, 95% CI 2-sided [-0.22 to 0.32], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Arm A vs Arm B; Statistical analysis at Week 10 based on comparison between treatment groups; Test type: Superiority or Other; p = 0.1255, Mixed Models Analysis; LS Mean Difference = 0.20, 95% CI 2-sided [-0.06 to 0.46], Standard Error of Mean 0.13

6. Secondary Outcome: Percentage of Participants With PGIC for Each Arm Compared at Week 5 (Visit 4) and at Week 10 (Visit 6)
Description: as for outcome 5
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
percentage of participants
  Week 5 - very much improved(n=84, 82) | 11.9 | 12.2
  Week 5 - much worse(n=84, 82) | 44.0 | 43.9
  Week 5 - much improved(n=84, 82) | 31.0 | 32.9
  Week 5 - minimally improved(n=84, 82) | 8.3 | 9.8
  Week 5 - no change(n=84, 82) | 4.8 | 1.2
  Week 5 - minimally worse(n=84, 82) | 0.0 | 0.0
  Week 5 - very much worse(n=84, 82) | 0.0 | 0.0
  Week 5 - missing(n=84, 82) | 0.0 | 0.0
  Week 10 - very much improved(n=81, 76) | 25.9 | 31.6
  Week 10 - much improved(n=81, 76) | 46.9 | 51.3
  Week 10 - minimally improved(n=81, 76) | 21.0 | 15.8
  Week 10 - no change(n=81, 76) | 4.9 | 0.0
  Week 10 - minimally worse(n=81, 76) | 0.0 | 1.3
  Week 10 - much worse(n=81, 76) | 1.2 | 0.0
  Week 10 - very much worse(n=81, 76) | 0.0 | 0.0
  Week 10 - missing(n=81, 76) | 0.0 | 0.0

7. Secondary Outcome: Change From Baseline in Weekly Mean of Daily Sleep Interference Rating Scale (SIRS) Compared Between Arms at Week 5 (Visit 4) and at Week 10 (Visit 6)
Description: The Daily Sleep Interference Rating Scale (SIRS) consists of an 11-point NRS ranging from 0 ("pain does not interfere with sleep") to 10 ("pain completely interferes with sleep" [unable to sleep due to pain]). Participants described how pain had interfered with their sleep during the past 24 hours: Select the number that best describes how your pain has interfered with your sleep during the past 24 hours on a scale from 0 to 10 where 0 represents 'does not interfere with sleep' and 10 represents 'completely interferes' which means you are unable to sleep due to pain.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5(n= 85, 79) | -2.46 (0.235) | -2.12 (0.236)
  Week 10(n=81, 75) | -3.69 (0.265) | -3.38 (0.268)
Statistical Analysis 1: Comparison: Arm A vs Arm B; Statistical analysis at Week 5 compared between treatment groups; Test type: Superiority or Other; p = 0.2856, Mixed Models Analysis; LS Mean Difference = -0.34, 95% CI 2-sided [-0.97 to 0.29], Standard Error of Mean 0.317
Statistical Analysis 2: Comparison: Arm A vs Arm B; Statistical analysis at Week 10 compared between treatment groups; Test type: Superiority or Other; p = 0.3987, Mixed Models Analysis; LS Mean Difference = -0.31, 95% CI 2-sided [-1.02 to 0.41], Standard Error of Mean 0.363

8. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS-A) Anxiety Scores at Week 5 (Visit 4) and Week 10 (Visit 6)
Description: The HADS is a self-administered questionnaire measuring anxiety. Each subscale consists of 7 statements and the participants respond as to how each item applies to them on a scale of 0 to 3 (0 = No anxiety, to 3 = Severe feelings of anxiety). Separate scores are calculated for each subscale and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score the more severe the anxiety.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5 (n=84, 82) | -2.23 (3.78) | -1.91 (3.23)
  Week 10 (n=81, 76) | -3.09 (4.34) | -2.68 (4.08)

9. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS-D) Depression Scores at Week 5 (Visit 4) and Week 10 (Visit 6)
Description: The HADS is a self-administered questionnaire measuring depression. Each subscale consists of 7 statements and the participants respond as to how each item applies to them on a scale of 0 to 3 (0 = No depression, to 3 = Severe feelings of depression). Separate scores are calculated for each subscale and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score the more severe the depression.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5 (n=84, 82) | -1.87 (4.18) | -1.35 (3.87)
  Week 10 (n=81, 76) | -2.57 (4.62) | -2.01 (3.84)

10. Secondary Outcome: Percentage of Days in Mild, Moderate and Severe Pain at Period 1 and Period 2
Description: Period 1 indicates from Visit 2 (baseline) to Visit 4 (Week 5). Period 2 indicates from Visit 4 (Week 5) to Visit 6 (Week 10). A rating of 0 is considered no pain; 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
Time Frame: Period 1 and Period 2
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
% of days
  Period 1 (n=88, 90) (Mild) | 19.1 (27.88) | 15.3 (28.13)
  Period 2 (n=84, 81) (Mild) | 33.5 (36.98) | 25.0 (34.50)
  Period 1 (n=88, 90) (Moderate) | 40.2 (34.07) | 37.6 (35.23)
  Period 2 (n=84, 81) (Moderate) | 33.2 (34.28) | 44.2 (39.41)
  Period 1 (n=88, 90) (Severe) | 38.8 (40.11) | 44.8 (40.76)
  Period 2 (n=84, 81) (Severe) | 26.5 (39.09) | 21.8 (34.91)

11. Secondary Outcome: Change From Baseline in Brief Pain Inventory Short Form (BPI sf) - Pain Severity Index Score at Week 5 and Week 10
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the past 24 hours. The Pain severity domain: The BPI severity domain includes pain at its 'worst,' 'least,' 'average,' and 'now' (current pain) on 0-10 NRS scales and takes the mean of these 4 items. Scores range from 0 (no pain) to 10 (pain as bad as you can imagine), therefore higher scores indicate greater pain severity.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5 (n=84, 82) | -1.75 (2.07) | -1.68 (1.86)
  Week 10 (n=81, 76) | -2.83 (2.26) | -2.99 (2.45)

12. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Sleep Disturbance Subscale at Week 5 and Week 10
Description: The MOS-Sleep Scale is a self-administered questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. With the exception of sleep adequacy, optimal sleep, and quantity, higher scores reflect greater impairment in the MOS-Sleep subscales. Sleep Disturbance: Range=0 to 100; higher scores indicate greater sleep disturbance. Negative changes indicate improvement.
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 91
Units on a scale
  Week 5 (n= 84, 82) | -21.3 (29.73) | -16.5 (25.92)
  Week 10 (n= 81, 76) | -27.1 (25.70) | -22.8 (25.04)

13. Secondary Outcome: Percentage of Participants With >= 30% Reduction From Baseline in the Weekly Mean Pain NRS Score at Week 5 and Week 10
Description: as for outcome 1
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 88 | 90
Percentage of participants
  Yes (Week 5) | 51.1 | 35.6
  No (Week 5) | 48.9 | 64.4
  Yes (Week 10) | 63.6 | 58.9
  No (Week 10) | 31.8 | 31.1

14. Secondary Outcome: Percentage of Participants With >= 50% Reduction From Baseline in the Weekly Mean Pain NRS Score at Week 5 and Week 10
Description: as for outcome 1
Time Frame: Week 5 and Week 10
Population: The FAS that comprised all participants who took at least one dose of study medication (either pregabalin or celecoxib).
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 88 | 90
Percentage of participants
  Yes (Week 5) | 25.0 | 20.0
  No (Week 5) | 75.0 | 80.0
  Yes (Week 10) | 42.0 | 37.8
  No (Week 10) | 53.4 | 52.2

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent throughout the study period including 28 calendar days after the last dose of study medication.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/89 | 2/91
Other Adverse Events (participants affected / at risk) | 28/89 | 19/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=89) | Arm B (N=91)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=89) | Arm B (N=91)
Dizziness (Nervous system disorders) | 12 | 12
Headache (Nervous system disorders) | 10 | 7
Somnolence (Nervous system disorders) | 12 | 7

LIMITATIONS AND CAVEATS:
The study was terminated as it had been determined that it was no longer operationally feasible to continue the trial. The study termination was not due to a safety issue or finding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.